CLINICAL TRIAL: NCT04136600
Title: A Study of EGFR Monoclonal Antibody (Cetuximab/Nimotuzumab) in Combination With Chemotherapy Compared With Chemotherapy Alone in Patients With EGFR-amplification Advanced Gastric Cancer
Brief Title: EGFR Monoclonal Antibody for Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Changzheng Hospital (Other)
Responsible Party: Principal Investigator, Yuan-Sheng Zang, Department Head, Shanghai Changzheng Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EGFR-GC
Record Dates: First submitted 2019-10-19; First posted 2019-10-23 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Gastric Cancer; Cetuximab; Nimotuzumab
MeSH Terms: conditions — Stomach Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EGFR antibody arm (Experimental): Participants received a dose of 500 mg/m2 Cetuximab iv on Day 1 of cycle every 3 weeks, or 400mg Nimotuzumab on Day 1 of cycle, every week, until disease progression. 12 cycles of mFOLFOX (5-fluorouracil (5-FU) 1,200 mg/m2/day for 46 hours, leucovorin 200 mg/m2, and oxaliplatin 85 mg/m2 biweekly). 6-8 cycles of CapOX (Xeloda, 1000 mg/m2 po twice daily for 14 days every 3 weeks + oxaliplatin 135mg/m2 every 3 weeks). 6-8 cycles of SOX (S-1, 60mg for BSA>1.5, 50 mg for 1.5>BSA>1.25 , 40mg for BSA<1.25 po twice daily for 14 days every 3 weeks + oxaliplatin 135mg/m2 every 3 weeks)
  Interventions: Drug: EGFR antibody and Chemotherapy
- Placebo arm (Placebo Comparator): 12 cycles of mFOLFOX (5-fluorouracil (5-FU) 1,200 mg/m2/day for 46 hours, leucovorin 200 mg/m2, and oxaliplatin 85 mg/m2 biweekly). 6-8 cycles of CapOX (Xeloda, 1000 mg/m2 po twice daily for 14 days every 3 weeks + oxaliplatin 135mg/m2 every 3 weeks). 6-8 cycles of SOX (S-1, 60mg for BSA>1.5, 50 mg for 1.5>BSA>1.25 , 40mg for BSA<1.25 po twice daily for 14 days every 3 weeks + oxaliplatin 135mg/m2 every 3 weeks)
  Interventions: Drug: Chemotherapy

INTERVENTIONS:
Drug: EGFR antibody and Chemotherapy — Drug: Cetuximab Cetuximab: 500 mg/m2 iv on Day 1 of cycle every 3 weeks, until disease progression.
  Other Names:
  Erbitux Drug: Nimotuzumab Nimotuzumab: 400mg iv on Day 1 of cycle, every week, until disease progression
  Drug: Fluoropyrimidine 5-fluorouracil (5-FU): 2,400 mg/m2/day iv in first 46 hours of cycle, every two weeks for 12 cycles
  Other Names:
  5-Fu Drug: Capecitabine Capecitabine: 1000 mg/m2 po twice daily for 14 days every 3 weeks, for 6 cycles
  Other Names:
  Xeloda Drug: S-1 S-1: 60mg for BSA>1.5, 50 mg for 1.5>BSA>1.25 , 40mg for BSA<1.25 po twice daily for 14 days every 3 weeks, for 6 cycles
  Other Names:
  S-1 Drug: Oxaliplatin Oxaliplatin: 85 mg/m2 iv on Day 1 of cycle, every 2 week for 12 cycles with 5-Fu; Oxaplatin: 130 mg/m2 iv on Day 1 of cycle, every 3 week for 6 cycles combined with S-1 or Capecitabine;
  Arms: EGFR antibody arm
Drug: Chemotherapy — Drug: Fluoropyrimidine 5-fluorouracil (5-FU): 2,400 mg/m2/day iv in first 46 hours of cycle, every two weeks for 12 cycles
  Other Names:
  5-Fu Drug: Capecitabine Capecitabine: 1000 mg/m2 po twice daily for 14 days every 3 weeks, for 6 cycles
  Other Names:
  Xeloda Drug: S-1 S-1: 60mg for BSA>1.5, 50 mg for 1.5>BSA>1.25 , 40mg for BSA<1.25 po twice daily for 14 days every 3 weeks, for 6 cycles
  Other Names:
  S-1 Drug: Oxaliplatin Oxaliplatin: 85 mg/m2 iv on Day 1 of cycle, every 2 week for 12 cycles with 5-Fu; Oxaplatin: 130 mg/m2 iv on Day 1 of cycle, every 3 week for 6 cycles combined with S-1 or Capecitabine;
  Arms: Placebo arm

SUMMARY:
This study is intended to evaluate efficacy and safety of EGFR monoclonal antibody (Cetuximab/Nimotuzumab) in combination with a chemotherapy in gastric cancer patients with EGFR amplification.

DETAILED DESCRIPTION:
This parallel, randomized, open-label, single-centre study will evaluate the effect on overall survival of EGFR monoclonal antibody (Cetuximab/Nimotuzumab) in combination with a chemotherapy compared to the chemotherapy alone in patients with EGFR-amplication advanced gastric cancer. Cetuximab will be administered as intravenous infusion of 500 mg/m2 (BSA) every 3 weeks, while nimotuzumab will be administered as intravenous infusion of 400mg every week. The chemotherapy consists of a combination of 12 cycles of mFOLFOX-6, 6-8 cycles of SOX, 6-8 cycles of CapOX. Treatment with cetuximab/nimotuzumab will continue until disease progression. The target sample size is 50-100 patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >=18 years of age
* Inoperable locally advanced, recurrent, and/or metastatic cancer of the stomach or gastro-esophageal junction Adenocarcinoma
* EGFR-Amplification tumors (Copy Number>=5 for tissue or blood Next Generation Sequence)
* Expected survival ≥ 3 month;
* ECOG / PS score: 0-2;
* the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min;

Exclusion Criteria:

* Previous chemotherapy for advanced/metastatic disease;
* Lack of physical integrity of the upper gastrointestinal tract, or malabsorption syndrome;
* History of cardiac disease;
* Dyspnoea at rest, due to complications of advanced malignancy or other disease, or patients who require supportive oxygen therapy;
* Patient can not comply with research program requirements or follow-up;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Evaluation of tumor burden until first documented progress through study completion, an average of 2 years
  Time from treatment beginning until disease progression
Objective Response Rate | Evaluation of tumor burden through study completion, an average of 2 years
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission.

SECONDARY OUTCOMES:
Overall Survival | From date of treatment beginning until the date of death from any cause through study completion, an average of 2 years
  Time from treatment beginning until death from any cause
Adverse Effect | Incidence of Treatment-related adverse Events through study completion, an average of 2 years
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medical Oncology, Shanghai Changzheng Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No